CLINICAL TRIAL: NCT02531347
Title: Treatment of Hypertension Using Telemedical Home Blood Pressure Measurements
Brief Title: Comparison of Telemedical and Conventional Treatment of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, Professor, Chief Physician, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20110013
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedical blood pressure monitoring (Experimental): Telemedical home blood pressure measurements for three days every second week. The average of all measures excluding day one is electronically transmitted to the General Practitioners. Following communication primarily by email or telephone.
  Interventions: Behavioral: Telemedical home blood pressure measurements
- Conventional blood pressure monitoring (Active Comparator): Conventional blood pressure monitoring
  Interventions: Behavioral: Conventional blood pressure monitoring

INTERVENTIONS:
Behavioral: Telemedical home blood pressure measurements
  Arms: Telemedical blood pressure monitoring
Behavioral: Conventional blood pressure monitoring
  Arms: Conventional blood pressure monitoring

SUMMARY:
The purpose of the study is to compare antihypertensive treatment based on either conventional blood pressure measurements or telemedical home blood pressure measurements.

Hypothesis is that telemedical treatment of hypertension is more effective in lowering blood pressure, is more cost-effective and provides better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 to 64 years
* Registered address in the Municipality of Holstebro
* Enrolment at a practice of one of the general practitioners who had agreed to participate in the study
* Telemedical home blood pressure measurement with ≥12 measurements on day 2 and 3.
* Elevated home blood pressure ≥135/85 (if diagnosed diabetes, chronic kidney disease or prior stroke ≥130/80)
* Hypertension confirmed by daytime ambulatory blood pressure ≥135/85 (if diagnosed diabetes, chronic kidney disease or prior stroke ≥130/80)
* ECG verified sinus rhythm

Exclusion Criteria:

* Unwillingness to participate
* Normotension
* Withdrawal of consent to participate

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 375 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction | 3 month
  Difference in daytime ambulatory blood pressure from baseline to followup between intervention and control group

SECONDARY OUTCOMES:
Number of patients reaching target blood pressure | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai Hoffmann-Petersen, MD, Principal Investigator — Department of Medical Research and Medicine, Holstebro Regional Hospital, Holstebro, Denmark

REFERENCES:
- [Derived] Hoffmann-Petersen N, Lauritzen T, Bech JN, Pedersen EB. Short-term telemedical home blood pressure monitoring does not improve blood pressure in uncomplicated hypertensive patients. J Hum Hypertens. 2017 Feb;31(2):93-98. doi: 10.1038/jhh.2016.43. Epub 2016 Jun 23. PMID 27334521